CLINICAL TRIAL: NCT03571945
Title: Impact of Bi-spectral Index Guided Inhalation Anaesthesia on the Incidence of Intraoperative Awareness in Indian Patient Population: A Prospective, Randomised, Multi-Centric Study
Brief Title: Incidence of Intraoperative Awareness in Indian Patient Population
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Coronavirus infection decrease in elective case list , also lack of response from other centers
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Consultant & Associate Professor, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EC/09/17/1253
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Intraoperative Awareness
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Intervention Model Description: 2000- patients aged 18-65 years scheduled for elective surgery under general anaesthesia will be randomly allocated to one of the following two groups:
  Group I [BIS Guided Group, n=1000]: GA will be monitored and controlled with Bi-spectral index (BIS).
  Group II [ETAG Guided Group, n=1000]: GA will be monitored and controlled with end-tidal anaesthesia gas concentration (ETAG).
Who Masked: Participant, Outcomes Assessor
Masking Description: The attending anaesthesiologist will not be blinded to the method of administering GA (BIS or ETAG guided) and recovery immediately after extubation inside the OR. However, the postoperative evaluation of intraoperative awareness and patient recovery profile will be evaluated by an independent assessor blinded to the technique of GA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BIS Guided Group (Active Comparator): GA will be monitored and controlled with Bi-spectral index (BIS) monitoring.The anaesthesiologist will be blinded to ETAG and MAC readings.
  Interventions: Device: Bi-spectral Index (BIS QUATRO REF #186-0106)
- ETAG Guided Group (Active Comparator): GA will be monitored and controlled with end-tidal anaesthesia gas (ETAG) monitoring.The anaesthesiologist will be blinded to the BIS readings.
  Interventions: Device: End tidal anaesthesia gas concentration (ETAG)

INTERVENTIONS:
Device: Bi-spectral Index (BIS QUATRO REF #186-0106) — GA will be monitored and controlled with Bi-spectral index (BIS).
  Arms: BIS Guided Group
Device: End tidal anaesthesia gas concentration (ETAG) — GA will be monitored and controlled with end-tidal anaesthesia gas concentration
  Arms: ETAG Guided Group

SUMMARY:
The profiling of bi-spectral index (BIS) monitored facilitation of general anesthesia (GA), including, anesthesia induction and maintenance of GA depth state, emergence characteristics, and postoperative recovery parameters, is now extensively available. However, majority of the data supporting the use of BIS have emanated from western Caucasian patient population. Though research on BIS monitoring have also emerged from Asian subcontinent, the data generated, at the best, is too scattered, random, and non-homogenous to reflect onto how BIS guidance fares in Asians on a population basis. We aim to undertake a multi-centric prospective cohort trial in Asian patient population to analyze as to whether BIS guidance toes the profiling and the evidence in Caucasians.

DETAILED DESCRIPTION:
After Institutional Ethics Committee approval and informed written patient consent, 2000 patients justifying inclusion and exclusion criteria ( will be included in this National, multi-centric, prospective, randomised, double-blind (patients, analyst), 2- arm trial.

All the patients scheduled for elective surgery under general anaesthesia will be randomly (simple computer generated random number table) allocated to one of the following two groups:

Group I [BIS Guided Group, n=1000]: GA will be monitored and controlled with Bi-spectral index (BIS).

Group II [ETAG Guided Group, n=1000]: GA will be monitored and controlled with end-tidal anaesthesia gas concentration (ETAG).

Sample Size Estimation To detect a difference in incidence of awareness of 0.04 % (a rate based on Mashour et al, Anesthesiology 2012) between the ETAG and BIS-guided group a total of 1800 patients will be required at a power of 80% with a type-II error 0f 0.5. To compensate for possible drop outs 10% additional patients will be recruited for the study. Therefore, the total sample size will include 2000 patients.

Randomization concealment: will be done using opaque sealed envelopes with alphabetic codes. In addition, before opening the envelope patient's data slip will be pasted on the envelopes.

Blinding: Investigator, assessor and the data analyst will be blinded to the method of GA (BIS or ETAG guided) Subgroup Analysis: Subgroup analysis will be specifically performed and reported if the data shows gender equivalence (i.e., at least 40% patients of either sex in each group).

Anaesthesia Technique:

Routine monitoring (EtCO2, pulse oximetery, EKG, NIBP) will be applied during the procedure. Anaesthesia will be induced with fentanyl 2-mcg/kg and propofol 1.5-2.5 mg/kg. Non-depolarizing muscle relaxant (vecuronium/ rocuronium/ atracurium) will be administered to facilitate tracheal intubation. GA will be maintained with inhalation regimen (sevoflurane/desflurane-oxygen-air mixture) to target age-related MAC range of 0.7 to 1.3. Corresponding BIS score and end-tidal agent concentration will be noted at 5-minute interval. While, in the BIS group the anaesthesiologist will be blinded to ETAG and MAC readings, in the ETAG group BIS display will be turned off. However, ETAG and MAC data will both be analyzed once the study is over. Although, the MAC will be titrated to haemodynamic goals (+20% baseline of SBP/MAP/Heart rate), it will be maintained within the prescribed range. On either side of the range of MAC, the haemodynamic depression/ activation will be responded to with vasopressor/vasodilators. At the end of surgery inhalation agent delivery will be stopped. The residual neuromuscular blockade will be reversed with neostigmine and glycopyrrolate.

The patients will be extubated once wide-awake and following commands. ASSESSMENT PARAMETERS Analysis of Intraoperative Awareness Quantitative: The participants will be subjected to modified Brice Interview 20 24-hours after surgery and after one month. The Brice interview at one month will be undertaken through telephonic contact and if awareness is present on any or both the occasions, a three-member independent awareness committee will review the incidence intensively. The awareness will be adjudicated in broad divisions, including, definite, possible, and no awareness. 21 No Awareness: No awareness or a perception of awareness that has a high probability of occurrence in the preoperative and the postoperative period.

Possible Awareness: There is a perception of awareness but the patient is unable to recall any event definitive indicative of awareness.

Definite Awareness: Perception of awareness that has clear recall or has a high likelihood of occurring in the intraoperative period.

Qualitative: After adjudication of a definite awareness by the awareness committee, the participants will be classified on the awareness pattern using the Michigan awareness classification instrument. 21 Class 1 will be defined by isolated auditory perception, Class 2 by tactile perceptions, Class 3 by pain experience, Class 4 by a feeling of paralysis and helplessness to move, and Class 5 by the presence of both paralysis and pain. If the awareness event is associated with distress the class will be modified with a suffix "D".

If definite awareness is present, the participants will be offered counselling sessions to ward off long-term behavioral changes and post-traumatic stress disorder (PTSD) The inter-reviewer observation will be analyzed for agreement using Fleiss's Kappa statistics for blinded assessment.

BIS score and end-tidal inhalation agent concentration: The intraoperative BIS scores and end-tidal inhalation agent concentration will be noted (every 5-minutes).

Time to awakening and tracheal extubation: Time (in minutes) to awakening will be noted after discontinuation of anaesthesia to point of first spontaneous eye opening. The time will be confirmed by the ability of the patient to obey commands. Time (in minutes) to tracheal extubation will comprise of the period after discontinuation of anaesthesia to tracheal extubation.

Statistical Analysis:

Demographic and procedural data will be analyzed with student's t-test, double sided, or the Chi-square test with Yate's correction as appropriate. Analysis of awareness outcome will be performed using Fisher's exact test. Sensitivity and specificity analysis will be undertaken for BIS values vis-à-vis explicit recall or no recall.

ELIGIBILITY:
Inclusion Criteria:

* Male or female gender
* Aged 18-65 yrs.
* ASA Physical Status I/II
* General Anaesthesia
* Elective Surgery
* Surgery duration > 30-minutes
* Consenting for follow-up

Exclusion Criteria:

* Uncompensated systemic co-morbidity
* Cardiac and Neurosurgical procedures
* Head & Neck surgery
* Obstetric surgery
* Emergency surgery
* Anticipated difficult airway
* H/O brain injury, EEG abnormality
* Neuropsychiatry disorders
* Substance abuse (opioids, alcohol, recreational drugs, benzodiazepine)
* Pacemakers & Electronic implants
* Obesity (BMI>30kg/m2)
* Adhesive allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2028-03-02 (Estimated); Study Completion 2028-03-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative awareness | From end of anaesthesia till 30-days postoperatively
  Will be assessed using Modified Brice Interview and Michigan awareness classification instrument

SECONDARY OUTCOMES:
Intraoperative Bi-spectral index (BIS) score | From beginning of anaesthesia (0-hours, baseline) till 8 hours intraoperatively
  BIS values will be recorded from the patient monitor
Intraoperative End-tidal anaesthesia gas (ETAG) concentration | From beginning of anaesthesia (0-hours, baseline) till 8 hours intraoperatively
  ETAG concentration will be recorded from the patient monitor
Intraoperative minimum alveolar concentration (MAC) | From beginning of anesthesia (0-hours, baseline) till 8 hours intraoperatively
  MAC will be recorded from the patient monitor
Recovery from anaesthesia | From end of anaesthesia till 20-minutes postoperatively
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Recovery from anaesthesia | From end of anaesthesia till 20-minutes postoperatively
  Time taken for tracheal extubation after discontinuation of anaesthesia will be noted
Changes in intra-operative heart rate (beats per minute) | From beginning of anesthesia (0-hours, baseline) till 8 hours intra-operatively
  Comparison of intra-operative heart rate between both the arms will be done
Change in Intra-operative blood pressure - systolic , diastolic, and mean (mmHg) | From beginning of anaesthesia (0-hours, baseline) till 8 hours intraoperatively]
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean between both the arms will be done
Postoperative Sedation | From end of anaesthesia till 24-hours postoperatively]
  Will be assessed using Modified Observer's assessment of alertness/sedation scale (OASS). This scale measures postoperative sedation on a scale of 0 to 5. A score of '0' indicates patient is deeply sedated with no response to any stimuli , whereas a score of 5 indicates that the patient is wide awake.
Postoperative Nausea and Vomiting (PONV) | From end of anaesthesia till 24-hours postoperatively]
  Will be assessed using postoperative nausea and vomiting (PONV) Scale. The scale measures PONV on a scale of 0 to 2. A score of '0' indicates that the patient has no emetic symptoms, whereas a score of '2' indicates that the patient has vomiting.
Postoperative Analgesia | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using 10-point Visual Analogue Scale (VAS) Score which measures pain on a scale of 0 to 10. A score of '0' indicates that the patient is free of pain whereas a score of '10' indicates that patient has severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Amitabh Dutta, MD, PhD, Study Chair — Sir Ganga Ram Hospital; Jayashree Sood, MD,FFRCA, Study Director — Sir Ganga Ram Hospital; Nitin Sethi, DNB, Principal Investigator — Sir Ganga Ram Hospital
Locations (5):
- India (5):
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Prof. L Parthasarathy, Chennai, Tamil Nadu
  - Post Graduate Institute For Medical Education & Research, Chandigarh
  - Apollo Gleneagles Hospital, Kolkata
  - P D Hinduja Hospital & Medical Research Centre, Mumbai

IPD SHARING:
Plan to Share IPD: Undecided